CLINICAL TRIAL: NCT07309549
Title: The Extended Study of Prevalence of Infection in Intensive Care IV (EPIC IV)
Brief Title: The Extended Study of Prevalence of Infection in Intensive Care IV
Acronym: EPIC IV
Status: Not yet recruiting | Type: Observational
Sponsor: Universidad de la Sabana (Other)
Collaborators: St. James's Hospital, Ireland (Other)
Responsible Party: Sponsor
Other Study IDs: Pending
Record Dates: First submitted 2025-12-15; First posted 2025-12-30 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Sepsis; Infection
Keywords: Intensive Care Unit; Critical Illness; Severe Infection; Organ Dysfunction; ICU Outcomes; Global Prevalence
MeSH Terms: conditions — Sepsis; Infections; Critical Illness

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- All patients present on or admitted to a contributing ICU on the study day: None interventions

SUMMARY:
The goal of this observational study is to learn how common infections are in intensive care units (ICUs) around the world and how they are treated. The study will look at all adults in the ICU during a single 24-hour period. The main questions it aims to answer are:

* What types of infections and antibiotic-resistant bacteria are most common in ICUs worldwide?
* How do resistance patterns affect how participants are treated and how they recover?

How are antibiotics used in ICUs, and how do hospitals practice antibiotic stewardship?

* What organ support treatments do participants with infections receive?
* What are the outcomes of participants with severe infections, including survival at hospital discharge (up to 60 days)?

Researchers will compare ICUs across regions and income levels to see how infection patterns, treatments, and outcomes differ around the world.

Participants will:

* Be counted if they are present in the ICU at any time during the study day.
* Have information collected from their medical record about their health, the infection they may have, treatments they receive, and their outcome at ICU and hospital discharge (up to 60 days).

Because this is an observational study, participants will not receive any new treatments as part of the study.

DETAILED DESCRIPTION:
The Extended Prevalence of Infection in Intensive Care IV (EPIC IV) study is an international, multicenter, prospective 24-hour point-prevalence study designed to provide an updated global assessment of infection patterns, antimicrobial use, organ support strategies, and related outcomes among adult patients treated in intensive care units (ICUs).

This study follows the methodology of previous EPIC initiatives (1998, 2007, 2017), while addressing the substantial changes in infection epidemiology observed in the post-COVID-19 era, including shifts in microbial resistance profiles and ICU practice patterns. Each participating ICU will select a single study day within the predefined window, during which all patients aged ≥18 years who are present in the unit at any time during the 24-hour period will be included.

Data collection will be standardized across sites and will include:

* Patient-level information on demographics, comorbidities, admission characteristics, severity-of-illness scores (APACHE II, SAPS II, SOFA), organ dysfunction, microbiology results, antimicrobial therapies, and supportive treatments.
* Unit-level characteristics related to ICU organization, staffing, resource availability, and antimicrobial stewardship practices.
* Follow-up data on ICU and hospital outcomes, censored at 60 days after the study day.

No study-specific treatments or interventions will be administered. All clinical care will follow local practice. Microbiological testing and therapeutic decisions will not be influenced by the study protocol.

EPIC IV will enable detailed analyses of global and regional variability in infection epidemiology, antimicrobial resistance, antibiotic stewardship performance, and resource utilization. The large international sample size will support predefined sub-studies examining associations between infection type, resistance patterns, comorbidities, ICU structural characteristics, and patient outcomes. The dataset will also allow stratified analyses based on country income level and geographical region, generating evidence relevant to both high-income and low- and middle-income countries.

This coordinated effort aims to produce a comprehensive and contemporary description of infectious disease burden in ICUs worldwide and to inform future clinical guidelines, policy development, and resource allocation.

ELIGIBILITY:
Inclusion Criteria:

* All adult patients (>18 years) treated in the participating ICUs on the study day.

Exclusion Criteria:

* Patients under 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A worldwide sample of adult patients who are present in participating intensive care units during a single 24-hour study period, regardless of diagnosis, treatment, or reason for ICU admission.
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2026-03 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
All-cause mortality at hospital discharge | Up to 60 days after the study day
  The primary outcome measure is all-cause mortality at hospital discharge, censored at 60 days from the study day. Mortality status will be assessed at ICU discharge and again at hospital discharge or Day 60, whichever occurs first.

SECONDARY OUTCOMES:
ICU mortality | From ICU admission to ICU discharge (up to 60 days)
  Proportion of enrolled patients who die during their stay in the Intensive Care Unit (ICU). Mortality will be assessed based on ICU discharge status and used to evaluate short-term outcomes among critically ill patients included in the study.
ICU and hospital lengths of stay | From ICU/hospital admission to discharge (up to 60 days)
  Duration of stay measured as the total number of days each patient spends in the ICU and the hospital, from admission until ICU and hospital discharge. These measures will be used to evaluate disease severity, resource utilization, and patient recovery patterns.
Organ Failure | From ICU/hospital admission to discharge (up to 60 days)
  Occurrence of new or worsening organ failure during ICU or hospital stay, assessed using validated clinical criteria (e.g., components of the SOFA score). Organ dysfunction will be evaluated to characterize severity of illness and its association with outcomes.
Antimicrobial Resistance | From ICU/hospital admission to discharge (up to 60 days)
  Presence and characterization of antimicrobial-resistant pathogens isolated from clinical specimens during ICU or hospital stay. Resistance will be defined according to standard microbiological and susceptibility testing methods and used to assess the burden and patterns of antimicrobial resistance across participating centers.

CONTACTS AND LOCATIONS:
Overall Officials: Ignacio-Martin Loeches, MD, PhD, FJFICMI, Principal Investigator — St James' Hospital. Dublin, Ireland; Luis Felipe Reyes, MD, MSc, PhD, Principal Investigator — Universidad de La Sabana. Chia, Colombia; Jean-Louis Vincent, MD, PhD, Principal Investigator — Erasme University Hospital. Brussels, Belgium

IPD SHARING:
Plan to Share IPD: Undecided
The decision regarding the sharing of individual participant data has not yet been finalized. IPD availability will depend on ethical approvals, institutional policies, and data-governance requirements across participating sites.

REFERENCES:
- [Background] Wynne C. Improve your children .... change yourself! Caritas. 1990 Autumn;56(75):11. No abstract available. PMID 2207816
- [Background] Vincent JL, Rello J, Marshall J, Silva E, Anzueto A, Martin CD, Moreno R, Lipman J, Gomersall C, Sakr Y, Reinhart K; EPIC II Group of Investigators. International study of the prevalence and outcomes of infection in intensive care units. JAMA. 2009 Dec 2;302(21):2323-9. doi: 10.1001/jama.2009.1754. PMID 19952319
- [Background] Vincent JL, Bihari DJ, Suter PM, Bruining HA, White J, Nicolas-Chanoin MH, Wolff M, Spencer RC, Hemmer M. The prevalence of nosocomial infection in intensive care units in Europe. Results of the European Prevalence of Infection in Intensive Care (EPIC) Study. EPIC International Advisory Committee. JAMA. 1995 Aug 23-30;274(8):639-44. PMID 7637145
- [Background] Finfer S, Bellomo R, Lipman J, French C, Dobb G, Myburgh J. Adult-population incidence of severe sepsis in Australian and New Zealand intensive care units. Intensive Care Med. 2004 Apr;30(4):589-96. doi: 10.1007/s00134-004-2157-0. Epub 2004 Feb 12. PMID 14963646
- [Background] Brun-Buisson C, Meshaka P, Pinton P, Vallet B; EPISEPSIS Study Group. EPISEPSIS: a reappraisal of the epidemiology and outcome of severe sepsis in French intensive care units. Intensive Care Med. 2004 Apr;30(4):580-8. doi: 10.1007/s00134-003-2121-4. Epub 2004 Mar 2. PMID 14997295
- [Background] Weycker D, Akhras KS, Edelsberg J, Angus DC, Oster G. Long-term mortality and medical care charges in patients with severe sepsis. Crit Care Med. 2003 Sep;31(9):2316-23. doi: 10.1097/01.CCM.0000085178.80226.0B. PMID 14501962
- [Background] Padkin A, Goldfrad C, Brady AR, Young D, Black N, Rowan K. Epidemiology of severe sepsis occurring in the first 24 hrs in intensive care units in England, Wales, and Northern Ireland. Crit Care Med. 2003 Sep;31(9):2332-8. doi: 10.1097/01.CCM.0000085141.75513.2B. PMID 14501964
- [Background] Alberti C, Brun-Buisson C, Burchardi H, Martin C, Goodman S, Artigas A, Sicignano A, Palazzo M, Moreno R, Boulme R, Lepage E, Le Gall R. Epidemiology of sepsis and infection in ICU patients from an international multicentre cohort study. Intensive Care Med. 2002 Feb;28(2):108-21. doi: 10.1007/s00134-001-1143-z. Epub 2001 Dec 4. PMID 11907653
- [Background] Martin GS, Mannino DM, Eaton S, Moss M. The epidemiology of sepsis in the United States from 1979 through 2000. N Engl J Med. 2003 Apr 17;348(16):1546-54. doi: 10.1056/NEJMoa022139. PMID 12700374
- [Background] Angus DC, Linde-Zwirble WT, Lidicker J, Clermont G, Carcillo J, Pinsky MR. Epidemiology of severe sepsis in the United States: analysis of incidence, outcome, and associated costs of care. Crit Care Med. 2001 Jul;29(7):1303-10. doi: 10.1097/00003246-200107000-00002. PMID 11445675